CLINICAL TRIAL: NCT01230346
Title: Intervention to Promote Uptake of Cancer Risk Counseling for Underserved Latinas
Brief Title: Culturally-Informed Counseling in Latinas at High Risk for Hereditary Breast or Ovarian Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 08237; NCI-2010-01998
Record Dates: First submitted 2010-09-22; First posted 2010-10-29 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: No Evidence of Disease; BRCA1 Syndrome; BRCA2 Syndrome; Hereditary Female Breast Carcinoma; Hereditary Ovarian Carcinoma
MeSH Terms: interventions — Counseling; Early Intervention, Educational; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (Experimental): Patients receive a culturally-informed adapted motivational interviewing telephone call.
  Interventions: Other: questionnaire administration; Other: survey administration; Other: counseling intervention; Other: educational intervention
- Arm II (Experimental): Patients participate in a controlled condition comprising a health habits intervention group.
  Interventions: Other: questionnaire administration; Other: survey administration; Other: counseling intervention
- Arm III (Active Comparator): Patients receive usual care comprising a standard scheduling phone call and proceed with normal GCRA process.
  Interventions: Other: questionnaire administration; Other: survey administration

INTERVENTIONS:
Other: questionnaire administration — Ancillary studies
Other: survey administration — Ancillary studies
Other: counseling intervention — Telephone intervention
  Other Names: counseling and communications studies
  Arms: Arm I; Arm II
Other: educational intervention — Telephone intervention
  Other Names: intervention, educational
  Arms: Arm I

SUMMARY:
This pilot clinical trial studies a culturally-informed counseling intervention in Latinas at high risk for hereditary breast or ovarian cancer. A culturally-informed counseling intervention may be an effective method to help people learn more about their cancer risk.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To conduct a randomized trial of a culturally-informed pre-genetic cancer risk assessment (GCRA) telephone intervention.

II. To evaluate the effect of the pre-GCRA intervention versus a time and attention control versus standard scheduling procedure alone (usual care) on levels of anxiety, perceived personal control and cancer genetics knowledge.

III. To explore patients' experiences with the pre-GCRA intervention through post-intervention telephone interviews.

SECONDARY OBJECTIVES:

I. To explore patients' perceived barriers to GCRA through no-show telephone interviews.

OUTLINE:

Patients are randomized to 1 of 3 treatment arms.

ARM I: Patients receive a culturally-informed adapted motivational interviewing telephone call.

ARM II: Patients participate in a controlled condition comprising a health habits intervention group.

ARM III: Patients receive usual care comprising a standard scheduling phone call and proceed with normal GCRA process. All patients are mailed standard new patient packets containing questionnaires on demographics and personal health history, and a family history form. All patients then undergo genetic cancer risk assessment.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have a personal history of hereditary breast or ovarian cancer; a subset of 60 women without a personal history of hereditary or ovarian cancer will be included in an exploratory subset analysis
* Meet NCCN criteria for consideration of genetic testing for hereditary breast cancer
* Willing to sign consent
* Pregnant women and women of child-bearing potential are eligible for participation in this study
* Women who report themselves to be of Latino or Hispanic ethnic background (defined as Spanish, Mexican, Central or South American, Cuban, Puerto Rican, Dominican, or other Hispanic origin)
* Women who are under- or uninsured and come from low-income communities
* Ability to understand English or Spanish

Exclusion Criteria:

* Previous participation in GCRA

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2010-09-03 (Actual); Primary Completion 2016-11-10 (Actual); Study Completion 2026-09-25 (Estimated)

PRIMARY OUTCOMES:
Effect of pre-GCRA intervention versus a time and attention control versus standard scheduling procedure alone (usual) on levels of anxiety, perceived personal control and cancer genetic knowledge | One week after genetic cancer risk assessment (GCRA)
  Tested using 3 x 3 repeated measures analysis of covariance (ANCOVA)s in which the within subjects variables are anxiety or perceived control, the between groups variable is group membership, and covariates include fatalism and other appropriate moderators.
Experiences with the pre-GCRA intervention through post-intervention telephone interviews | One week after genetic cancer risk assessment (GCRA)
Conduct a randomized controlled trial of a culturally-informed pre-GCRA telephone intervention utilizing AMI techniques | One week after genetic cancer risk assessment (GCRA)
  Will use a multivariate ANCOVA (MANCOVA) to test for group differences among all five preparedness scores, with step-down F ratios of each individual score, using fatalism and other moderators as covariates, as appropriate.

SECONDARY OUTCOMES:
Perceived barriers to GCRA through no-show telephone interviews | One week after genetic cancer risk assessment (GCRA)

CONTACTS AND LOCATIONS:
Overall Officials: Bita Nehoray, Principal Investigator — City of Hope Medical Center
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - University of Southern California-Keck School of Medicine, Los Angeles, California
  - Olive View-UCLA Medical Center, Sylmar, California